CLINICAL TRIAL: NCT03732170
Title: Clinical Outcome of Root Canal Treatment With TotalFill® Bioceramic Sealer and AH Plus® Sealer: A Randomized Controlled Trial
Brief Title: Root Canal Treatment With TotalFill® Bioceramic Sealer and AH Plus® Sealer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018/00390
Record Dates: First submitted 2018-11-01; First posted 2018-11-06 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Root Canal Obturation

STUDY DESIGN:
Intervention Model Description: Study subject (tooth) will be randomized in a 1:1 allocation ratio between the two treatment groups.
Who Masked: Participant, Outcomes Assessor
Masking Description: Blinding will be done to the assessors to reduce bias to healing assessment. As well, participants won't know which treatment they are undergoing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TotalFill® Bioceramic sealer (Experimental): It will be used in conjunction with TotalFill® bioceramic impregnated gutta percha points for the obturation of root canals. It is dispensed through a fine disposable syringe into the root canals during obturation.
  Interventions: Device: TotalFill® Bioceramic sealer
- AH plus® sealer (Active Comparator): It consists of 2 pastes that are mixed together in equal amounts before it is used in conjunction with gutta percha points for obturation during root canal treatment.
  Interventions: Device: AH plus® sealer

INTERVENTIONS:
Device: TotalFill® Bioceramic sealer — The participant will be treated with TotalFill® Bioceramic sealer.
  Arms: TotalFill® Bioceramic sealer
Device: AH plus® sealer — The participant will be treated with AH plus® sealer.
  Arms: AH plus® sealer

SUMMARY:
The study design is a double blinded randomized controlled trial and 170 subjects (teeth) , 85 in each of the 2 groups, will be enrolled from the patients at the NUH dental centre endodontic unit. The study aims to assess how the use of TotalFill® bioceramic sealer affects the healing outcome of apical periodontitis compared to a control AH plus®.

Conventional root canal treatment will be done during this study. Radiographs will be taken at each study visit during the study for root canal. The preoperative, postoperative and review clinical and radiographic data will be analysed.

DETAILED DESCRIPTION:
Randomization and Blinding Study subject (tooth) will be randomized in a 1:1 allocation ratio between the two treatment groups. Allocation will be by random permuted block and stratified by gender to enhance balance. Computer generated randomized allocation for each subject will be concealed in opaque envelope. The envelope will only be opened by the operator on the obturation visit of the enrolled patient and the randomization number assigned to them.

In the event that a patient has more than 1 tooth eligible for the study, only one tooth on left and/or right side of the mouth will be recruited for the study. Therefore, a patient could contribute a maximum of two teeth for this study (i.e. a maximum of one tooth on each side of the mouth). Selection of tooth will be done using computer generated randomization number.

Study Visits and Procedures After cleaning and shaping and the patients are deemed ready for obturation, the patients will be randomly assigned to one of the 2 groups for obturation using AH plus® or TotalFill® bioceramic sealer.

* The patients and the examiners will be blinded to the type of sealer used but it would not be possible to blind the operators.

  b. Post Study Follow up and Procedures
* A follow up phone call will be made to collect the patient pain experience on day 1, day 3 and day 7 post treatment which they have recorded on their pain/discomfort diary.
* At the 6-month and 12-month review, patients will be examined for any clinical signs and symptoms and a review radiograph will be taken to assess the size of the periapical lesion.

  c. Radiographic assessment
* All radiographs will be taken with a localising device to control for angulation and magnification.
* Calibrated measurement tools in the dental practice management software will be used to measure the diameter of the lesion across the longest diameter.

Statistical and Analytical Plans

a. General Considerations Intention-to-treat population is considered the main analysis population. The intention-to-treat population includes all subjects who were assigned a randomization number. Study subject's demographic and pre-operative characteristics will be summarized for each treatment group.

ELIGIBILITY:
Inclusion Criteria:

* A preoperative periapical radiograph will be required for diagnosis.
* Subjects at least 21 years old.
* Medically healthy
* In a patient with multiple teeth requiring root canal treatment, only 1 tooth from each side will be included and selected at random.

Exclusion Criteria:

* Patient below 21 years old
* Pregnant women.
* Patients with autoimmune diseases and uncontrolled diabetes.
* Teeth with periodontal probing depths of 5mm or more.
* Incomplete root formation that is detected radiographically.
* Cracked teeth
* Teeth are deemed to have poor restorative prognosis.
* Teeth with adjacent teeth on the same side that require root canal treatment

Ages: 21 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2018-08-13 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in the status of periapical lesion size | comparison of the periapical lesion size at baseline, 6 month and 12 month
  Proportion z-test will be carried to compare the proportion of study subjects with improved apical lesion size between the two treatment groups. Odds ratio with 95% confidence interval will be reported. Logistic regression analysis adjusted for the stratification variables (gender) and other confounding factors (namely patency, extrusion of sealer or GP, short fill, voids, pre-op apical size, pre-op clinical symptoms and number of C&S visits).

SECONDARY OUTCOMES:
Comparison of the pain score of post-op pain | Day 1, Day 3 and Day 7 post treatment
  Proportion z-test will be carried out. The odds ratio with a 95% confidence interval will be reported. A two-sample t-test will be performed to access the change in pain score (Pain was recorded as "no pain" (score = 0) or a 5-point Likert scale ranging from very mild pain (score = 1) to severe pain (score = 5)) at post-op compared with pre-op between the two treatment groups. Shapiro Wilk's test and Levene's test will be performed to check the normality and homogenous variance assumption of the two-sample t-test. Non-parametric approach (Mann-Whitney U-test) will be employed if there is significant violations of the normality assumption.

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Yu, PhD, Principal Investigator — National University Hosptial, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP